CLINICAL TRIAL: NCT04456478
Title: Randomized Trial in Assisted Reproductive Technology : Impact of PH Values of the Embryo Culture Medium on Live Birth Rate After in Vitro Fertilization (IVF)
Brief Title: Impact of PH Values of the Embryo Culture Medium on Success of in Vitro Fertilization (IVF)
Acronym: ACIDOFIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RC31/19/0503; 2020-A00221-38 (Other: ID RCB)
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Embryo Growth Disorder; Humans; Pregnancy
Keywords: pH; embryo culture; In Vitro Fertilization; live birth rate; randomized trial

STUDY DESIGN:
Intervention Model Description: Multicentric randomized blinded trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pH 7.38 ± 0.02 (Active Comparator): IVF-ICSI will be performed according to the usual procedure and the day of the oocyte puncture, the embryologist will proceed to the culture of the oocytes and embryos in the culture medium with a pH at 7.38 ± 0.02
  Interventions: Procedure: pH at 7.38 ± 0.02
- pH 7.22 ± 0.02 (Experimental): IVF-ICSI will be performed according to the usual procedure and the day of the oocyte puncture, the embryologist will proceed to the culture of the oocytes and embryos in the culture medium with a pH at 7.22 ± 0.02
  Interventions: Procedure: pH at 7.22 ± 0.02

INTERVENTIONS:
Procedure: pH at 7.38 ± 0.02 — In the 3 centers of the study, IVF-ICSI will be performed according to the usual procedure: ovarian stimulation, oocyte retrieval, sperm microinjection by ICSI, embryo culture in Global® Total HSA medium, embryo selection and transfer at day 3. The day of the oocyte puncture, the embryologist will proceed to the 1: 1 randomization: culture of the embryos in a medium with a pH at 7.38 ± 0.02. We have chosen to study specifically the early stages of fertilization and embryo development (until day 3), stages for which extracellular pH control is more critical because the intracellular pH regulatory mechanisms are somewhat limited and could be exceeded.
  Arms: pH 7.38 ± 0.02
Procedure: pH at 7.22 ± 0.02 — In the 3 centers of the study, IVF-ICSI will be performed according to the usual procedure: ovarian stimulation, oocyte retrieval, sperm microinjection by ICSI, embryo culture in Global® Total HSA medium, embryo selection and transfer at day 3. The day of the oocyte puncture, the embryologist will proceed to the 1: 1 randomization: culture of the embryos in a medium with a pH at 7.22 ± 0.02. We have chosen to study specifically the early stages of fertilization and embryo development (until day 3), stages for which extracellular pH control is more critical because the intracellular pH regulatory mechanisms are somewhat limited and could be exceeded.
  Arms: pH 7.22 ± 0.02

SUMMARY:
The objective of this study is to compare, through a multicentric randomized trial, the impact of two pH values in the embryo culture medium on the clinical results of In Vitro Fertilization (IVF) process and especially the impact on live birth delivery rate.

DETAILED DESCRIPTION:
Despite progress in Assisted Reproductive Technology (ART), the livebirth rate per oocyte retrieval during In Vitro Fertilization (IVF) remain relatively low (15 à 25%). This is in part due to the sensitivity of the preimplantation embryo to its environment. Indeed, there is growing evidence that culture conditions during IVF are critical not only for the development of pre- and post-implantation embryo, but also for long-term health effects; and numerous animal data suggest the importance of pH control in the IVF culture medium. Maintaining the intercellular pH (pHi) is one of the vital roles of embryo homeostasis since pHi regulates many cellular processes. Indeed, variations in pHi can affect embryonic development. Although the embryo has biochemical systems to regulate its pHi, these systems can be overtaken. Under the conditions of IVF embryo culture, the extracellular pH (pHe) in a culture medium is the result of a balance between CO2 concentration in the incubator and bicarbonate concentration in the culture medium (determined by the medium manufacturer). The recommendations of the manufacturers of embryo culture media are to maintain a pHe slightly higher (generally between 7.2 and 7.4) than the pHi (estimated between 7.1 to 7.2) to compensate for the acidification due to cell metabolism. However, as the pH scale is logarithmic, a pHe variation of 7.2 to 7.4 corresponds to a decrease in the concentration of H+ ions by a factor of 1.6 in the medium. Actually, there is no clinical data to know what is the ideal pH to apply to a culture medium during IVF.

This is a clinical study comparing two pH values in the culture medium of embryos obtained by IVF, randomized, multicentric (3 centers), patient-blinded, in groups parallel to the ratio 1: 1. IVF-ICSI will be performed according to the usual procedure and the day of the oocyte puncture, the embryologist will proceed to the 1: 1 randomization: culture of the oocytes and embryos in the culture medium with a pH at 7.38 ± 0.02 or a pH at 7.22 ± 0.02.

In case of pregnancy after embryo transfer, patients will be followed until delivery.

ELIGIBILITY:
Inclusion Criteria:

* Couples whose woman is 18 to 40 years old and man is 18 to 60 at the time of inclusion.
* Infertile couple with a medical indication of IVF-ICSI according to criteria applied in each center.
* First or second ICSI attempt with fresh embryo transfer.
* Signature of informed consent by both partners of the couple
* Affiliation to a social security scheme or equivalent for both partners of the couple.
* Fitting the inclusion criteria for IVF according the the French law.

Exclusion Criteria:

* Use of spermatozoa extracted by testicular biopsy.
* Freeze-al strategy (without fresh embryo transfer) decided before embryo culture
* Absence of mature oocyte (metaphase II) at the day of the puncture
* Uterine pathology affecting implantation (uterine malformation, diffuse adenomyosis ...)
* One of the two partners (or both) is (are) infected with HIV, HCV or HBV in the year before the inclusion
* One of the two partners (or both) is (are) in safeguarding justice, under guardianship or trusteeship.
* Couple having already participated once in the study.
* Couple enrolled in another interventional clinical study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Couples whose woman is 18 to 40 years old and man is 18 to 60 at the time of inclusion because the study concerns in vitro fertilization
Enrollment: 429 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Live birth delivery rate | month 9
  Number of deliveries that resulted in at least one live birth (gestational age ≥ 22 weeks) / Number of oocyte retrievals

SECONDARY OUTCOMES:
Fertilization rate | day 1
  Number of 2PN zygotes at day 1 post-injection / Number of matures injected oocytes
Cleavage rate | day 2
  Number of embryos with at least 2 blastomeres at day 2 / Number of diploid zygotes at day 1 post-injection
Percentage of top embryos | day 3
  Number of 7 to 10-blastomeres embryos at day 3 with less than 10% fragments / Total number of embryos at day 3
Embryo freezing rate | day 6
  Number of frozen embryos / Total number of obtained embryos
Implantation rate | week 5
  Number of gestational sacs observed with ultrasonography (5 weeks after embryo transfer) divided by the number of embryos transferred (expressed as a percentage)
Clinical ongoing pregnancy rate by transfer | week 5
  Number of pregnancies diagnosed by ultrasonographic of at least one fetus with a discernible heartbeat at 5 weeks after embryo transfer / Number of embryo transfers
Clinical ongoing pregnancy rate by oocyte retrieval | week 5
  Number of pregnancies diagnosed by ultrasonographic of at least one fetus with a discernible heartbeat at 5 weeks after embryo transfer / Number of oocyte retrieval
Miscarriage rate | week 22
  Number of spontaneous loss of an intrauterine pregnancy prior to 22 completed weeks of gestational age / Number of pregnancies
Malformation rate diagnosed at birth | month 9
  Number of malformations according to Eurocat classification (in total and in Eurocat subgroups) / Total number of newborns

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GATIMEL, ph, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - CHU de BORDEAUX, Bordeaux
  - Centre AMP BIOPYRENEES, Pau
  - CHU de TOULOUSE, Toulouse